CLINICAL TRIAL: NCT02578420
Title: Back to Basics - Effects, Narratives and Routes of Administration of Open-label Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EKNZ 2015-246
Record Dates: First submitted 2015-10-12; First posted 2015-10-19 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Placebo Effect; Pain; Expectancy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- open-label placebo (Placebo Comparator): Participants (N=40) will have the information that they are receiving an inert cream (i.e. "placebo"). Placebo will be described as an inert or inactive cream, with no medication in it. Additionally, participants will be told that "placebo has been shown in rigorous clinical testing to produce significant mind-body self-healing processes." The placebo administration will be combined with the following scientific rationale/verbal suggestion: (a) placebos are effective analgesics, (b) classical conditioning as a possible mechanism of this effect, (c) compliance is important for outcome and (d) positive expectations increase placebo effects, but are not necessary.
  Interventions: Other: open-label placebo
- deceptive placebo (Sham Comparator): Participants (N=40) will have the information that they are receiving an analgesic cream ("Antidolor, containing "Lidocain"), while in fact they will receive an inert cream, only. Antidolor will be described as an analgesic cream.
  Interventions: Other: deceptive placebo
- control group (Placebo Comparator): Participants (N=40) will have the information that they are receiving an inert control cream.
  Interventions: Other: open-label placebo
- no treatment group (No Intervention): Participants (N=40) will be told that they are in the "no treatment group" and that they will not receive an analgesic cream.

INTERVENTIONS:
Other: open-label placebo — Placebo Cream, openly described as "Placebo"
  Arms: control group; open-label placebo
Other: deceptive placebo — Placebo Cream, described as "Voltaren, containing Diclofenac"
  Arms: deceptive placebo

SUMMARY:
To date, very little is known about the mechanisms of open-label placebo treatment and there is a lack in highly controlled experimental designs. Therefore, the planned project will test well-established explanatory models of (deceptive) placebo, i.e., (1) expectancy, (2) meaning response, in an open-label placebo design, investigating their influence on placebo analgesia.

DETAILED DESCRIPTION:
The current project will consist of one experimental study and one qualitative study:

1. the effects of open-label, and deceptive placebo administration on placebo analgesia will be directly compared when both groups have a comparable expectancy-inducing scientific rationale;
2. subjective meaning models will be assessed by comparing subjective narratives of the placebo effect in open-label and deceptive placebo groups in a nested qualitative study.

The experimental study will be a randomized experiment with healthy subjects (N=120), and pain will be induced using a standardized heat pain paradigm (Medoc, Ramatishai, Israel; thermo-sensory analyzer (TSA)-II). Effects of the experimental conditions will be assessed both objectively (i.e. heat pain threshold and tolerance) and subjectively (i.e. subjective pain ratings, pain intensity and unpleasantness). Furthermore, investigators will randomly select 30 participants to take part in a nested qualitative study in order to qualitatively assess the meaning response by comparing subjective narratives of the placebo effect in the open-label and deceptive placebo groups, as well as in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults aged 18-65
* Healthy by self-report statement, thus no known current or chronic somatic diseases or psychiatric disorders
* Right-handedness (Oldfield, 1971),
* Willing to participate in study

Exclusion Criteria:

* Medicine or Psychology Students
* Any acute or chronic disease (chronic pain, hypertension, heart disease, renal disease, liver disease, diabetes) as well as skin pathologies, neuropathies or nerve entrapment symptoms, sensory abnormalities affecting the tactile or thermal modality
* Current medications (psychoactive medication, narcotics, intake of analgesics) or being currently in psychological or psychiatric treatment
* Insufficient German language skills to understand the instructions
* Previous participation in studies using pain assessment (threshold and tolerance) with Peltier Devices
* Daily consumption of more than three alcoholic standard beverages per day (a standard alcoholic beverage is defined as either 3dl beer or 1 dl wine or 2cl spirits)
* Current or regular drug consumption (THC, cocaine, heroin, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01; Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
subjective intensity and unpleasantness ratings of heat pain tolerance | 2 hours
  Visual Analogue Scale (VAS)
objective heat pain tolerance | 2 hours
  Temperatures

SECONDARY OUTCOMES:
Expectancy of Relief Scale (ERS; Erwartungsfragebogen) | 2 hours
Credibility and Effectiveness of the placebo analgesia expectation; adapted Version of the Context Model Questionnaire; Kontextmodellfragebogen (KMF) | 2 hours
multidimensional sensitivities questionnaire (Mehrdimensionaler Befindlichkeitsfragebogen (MDBF)) | 2 hours
sociodemographic questionnaire (Soziodemographischer Fragebogen (SDD)) | 2 hours
Revised Life Orientation Test (LOT-R) | 2 hours
NEO five-factor inventory (NEO-FFI) | 2 hours
questionnaire on competence and locus of control (Fragebogen zu Kompetenz- und Kontrollüberzeugungen (FKK)) | 2 hours
Anxiety and Depression Scale (HADS-D) | 2 hours
Beliefs in holistic health and holistic treatments; Complementary and Alternative Medicine Beliefs Intentory (CAMBI) | 2 hours
Desire for Relief Scale (DRS) | 2 hours
subjective intensity and unpleasantness ratings of heat pain threshold | 2 hours
  Visual Analogue Scale (VAS)
objective heat pain threshold | 2 hours
  Temperatures

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gaab, Prof, Study Chair — Clinical Psychology and Psychotherapy, Department of Psychology, University of Basel
Locations (1):
- University of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Locher C, Buergler S, Frey Nascimento A, Kost L, Blease C, Gaab J. Lay perspectives of the open-label placebo rationale: a qualitative study of participants in an experimental trial. BMJ Open. 2021 Aug 18;11(8):e053346. doi: 10.1136/bmjopen-2021-053346. PMID 34408060